CLINICAL TRIAL: NCT06405906
Title: Rationale Diet for Gallstone Disease (RADIGAL Trial): A Randomized Controlled Trial Comparing Fat-free Versus Balanced (WHO) Diet in Gallstone Disease
Brief Title: A Randomized Controlled Trial Comparing Fat-free Versus Balanced (WHO) Diet in Gallstone Disease
Acronym: RADIGAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Crete (Other)
Responsible Party: Principal Investigator, Konstantinos Lasithiotakis, Assistant Professor of Surgery, University Hospital of Crete
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 5414/27-03-2024
Record Dates: First submitted 2024-05-04; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Gallstone Disease; Gallstone; Colic; Gallstone; Cholecystitis, Acute; Cholelithiases; Postcholecystectomy Syndrome; Dietary Habits
Keywords: gallstone disease; cholecystitis; cholecystectomy; gallbladder diet
MeSH Terms: conditions — Cholelithiasis; Gallstones; Colic; Cholecystitis; Postcholecystectomy Syndrome; Feeding Behavior | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Biliary Colic Group - Non-operative Treatment - RADIGAL1 (Experimental): Patients presenting with biliary colic and treated non-operatively will be randomly assigned to receive fat-free diet or balanced WHO diet for 3 months.
  Interventions: Other: Fat-free diet; Other: Balanced WHO diet
- Cholecystitis Group - Non-operative Treatment - RADIGAL1 (Experimental): Patients presenting with acute cholecystitis and treated non-operatively will be randomly assigned to receive fat-free diet or balanced WHO diet for 3 months.
  Interventions: Other: Fat-free diet; Other: Balanced WHO diet
- Biliary Colic Group - Cholecystectomy - RADIGAL2 (Experimental): Patients undergoing cholecystectomy due to biliary colic will be randomly assigned to receive fat-free diet or balanced diet for 3 months.
  Interventions: Other: Fat-free diet; Other: Balanced WHO diet
- Cholecystitis Group - Cholecystectomy - RADIGAL2 (Experimental): Patients undergoing cholecystectomy due to acute cholecystitis will be randomly assigned to receive fat-free diet or balanced diet for 3 months.
  Interventions: Other: Fat-free diet; Other: Balanced WHO diet

INTERVENTIONS:
Other: Fat-free diet — The low-fat diet will consist of instructions to avoid fatty foods.
Other: Balanced WHO diet — The balanced WHO diet will adhere to the recommendations of the World Health Organization (WHO) and the Dietary Guidelines for Americans 2020-2025

SUMMARY:
The goal of this trial is to assess the effect on the quality of life (QoL) of recommending a fat-free diet versus a balanced WHO diet in symptomatic patients with gallstones and in patients undergoing cholecystectomy for gallstone disease. The main question it aims to answer is:

• Is balanced WHO diet as good as low-fat diet in terms of patient reported outcomes when gallstone disease is managed non-operatively (RADIGAL-1) or cholecystectomy is performed (RADIGAL-2)?

A validated QoL questionnaire (Gastrointestinal Quality of Life Index - GIQLI) will be administered both at baseline and during follow-up. Analysis of covariance with ordinary least squares estimation will be applied to estimate between-group differences in GIQLI scores at 3 months (primary endpoint). Patient adherence and the disease-related symptoms occurrence or hospitalizations will also be appraised (secondary endpoint).

Participants presenting with biliary colic or acute cholecystitis (RADIGAL-1) or undergoing cholecystectomy for gallstones (RADIGAL-2) will:

* be randomly assigned to recommending either a fat-free or a balanced WHO diet .
* be contacted via phone call to complete the GIQLI questionnaire and document overall adherence to the diets and secondary outcome events.

This trial examines the impact of diet on adverse events in gallstone disease, representing the first randomized study to focus on this aspect.

ELIGIBILITY:
Inclusion Criteria (RADIGAL1):

* 18 years old or older
* presenting with biliary colic in the ED or outpatient clinic, with the surgical team deciding to proceed with non-operative treatment (Group 1)
* presenting with acute calculous cholecystitis in the ED, with the surgical team deciding to proceed with non-operative management (Group 2)

Exclusion Criteria (RADIGAL1):

* history of gastrointestinal disease which might affect diet, e.g., inflammatory bowel disease, irritable bowel syndrome, short bowel syndrome
* inability to provide informed consent
* unwillingness to adhere to the recommended diet
* food allergies or intolerances that would prevent following the diet
* dietary habits (e.g., vegetarians, vegans) that preclude adherence to the recommended diet
* gallstone related cholangitis without biliary colic or cholecystitis
* complications from acute pancreatitis, such as pseudocysts, walled off necrosis, among others

Inclusion Criteria (RADIGAL2):

* 18 years old or older
* undergoing uncomplicated cholecystectomy (open or laparoscopic without bile duct exploration) due to a history of biliary colic (Group 1)
* undergoing uncomplicated cholecystectomy (open or laparoscopic without bile duct exploration) due to acute cholecystitis (Group 2)

Exclusion Criteria (RADIGAL2):

* history of gastrointestinal disease which might affect diet, e.g., inflammatory bowel disease, irritable bowel syndrome, short bowel syndrome
* inability to provide informed consent
* unwillingness to adhere to the recommended diet
* food allergies or intolerances that would prevent following the diet - dietary habits (e.g., vegetarians, vegans) that preclude adherence to the recommended diet
* gallstone related cholangitis without biliary colic or cholecystitis
* complications from acute pancreatitis, such as pseudocysts, walled off necrosis, among others
* choledocholithiasis
* complicated cholecystectomy
* patients undergoing subtotal cholecystectomy
* whether primary operation differs from cholecystectomy (e.g., colectomy)
* patients having treated with percutaneous cholecystostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life as measured by the GIQLI score (RADIGAL1/2) | Baseline, 3-month follow-up
  The GIQLI questionnaire contains 36 questions on gastrointestinal symptoms (19 items), physical status (7 items), emotional status (5 items), and social function status (5 items). Patient responses are recorded as 'all the time, most of the time, some of the time, a little of the time, or never'. The most favorable option is scored as 4 points, whereas the least favorable option receives 0 points.

SECONDARY OUTCOMES:
Patient adherence to the suggested diet (RADIGAL1/2) | Baseline, 3-month follow-up
  Patients will be queried if they followed the given diet daily, more than half the days of the month, less than half the days of the month or not at all.
Unplanned Emergency Department (ED) visit or hospital admission (RADIGAL1/2) | Baseline, 3-month follow-up
  Patients will be asked about emergency department visits or hospital admissions related to the gallstone disease.
Symptom Recurrence (RADIGAL1/2) | Baseline, 3-month follow-up
  Patients will be asked if they experienced postprandial abdominal pain, nausea, vomiting, or dyspepsia.
Unplanned or elective cholecystectomy (RADIGAL1) | Baseline, 3-month follow-up
  Patients who treated non-operatively will be asked if they underwent unplanned or elective surgery.
Time of Diet Discontinuation (weeks or months) (RADIGAL1/2) | Baseline, 3-month follow-up
  Patients will be asked how long after the first visit or discharge they stopped following the given diet.
Reason for discontinuing diet (RADIGAL1/2) | Baseline, 3-month follow-up
  Patients will be asked if the reason for discontinuing the given diet is one of the following: Improvement or absence of symptoms
  * No improvement of symptoms
  * Worsening of symptoms
  * Personal reasons
  * Inability to adhere to the diet for such a long period
  * Hospital admission
  * Advice from another surgeon.
Food categories chosen when not following diet (RADIGAL1/2) | Baseline, 3-month follow-up
  Patients will be asked which of the following food categories they chose to consume when they stopped following the suggested diet:
  * Fatty and red meats
  * Fried and butter products
  * Sugar, soft drinks, sweets, and processed snacks
  * Fatty dairy products
  * High salt and cold cuts

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Lasithiotakis, MD, PhD, Principal Investigator — Department of Surgery, University Hospital of Heraklion
Locations (1):
- Department of Surgery, University Hospital of Heraklion, Heraklion, Greece

IPD SHARING:
Plan to Share IPD: No